CLINICAL TRIAL: NCT06487988
Title: Asleep Fiberoptic vs Direct Laryngoscopy Effect on Hemodynamic Stability Using Opioid Free Anesthesia Induction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Christian Rouphael, Clinical Instructor of Anesthesia, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BIO-2023-0271
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Analgesics, Opioid; Anesthesia, General; Heart Rate; Blood Pressure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The direct conventional laryngoscopy group (Active Comparator): The direct conventional laryngoscopy group will be performed with N3 (for females) or N4 (for males) Macintosh laryngoscope blade.
  Interventions: Device: direct conventional laryngoscopy
- The fiberoptic guided intubation group (Experimental): The fiberoptic guided intubation will be performed.
  Interventions: Device: fiberoptic guided intubation

INTERVENTIONS:
Device: direct conventional laryngoscopy — direct conventional laryngoscopy will be performed with N3 (for females) or N4 (for males) Macintosh laryngoscope blade.
  Arms: The direct conventional laryngoscopy group
Device: fiberoptic guided intubation — fiberoptic guided intubation will be performed.
  Arms: The fiberoptic guided intubation group

SUMMARY:
The goal of this clinical trial is to compare blood pressure and heart rate between the fiberoptic and direct oral intubation using opioid free anesthesia induction. Secondary objectives include comparing the time needed for intubation and the incidence of postoperative sore throat, hoarseness, and upper airway trauma in adults aging between 18 to 55 years, scheduled for elective surgery under general anesthesia.

The main question it aims to answer is:

Does fiberoptic intubation cause less hemodynamic instability than direct oral intubation using opioid free anesthesia induction?

DETAILED DESCRIPTION:
Background: Intubation has always been linked to a transient increase in blood pressure and heart rate that could be deleterious in elderly and hemodynamically unstable patients. Fiberoptic intubation, which is currently used for suspected difficult intubation, could cause less marked rise in blood pressure and heart rate. Furthermore, "opioid free anesthesia" has gained popularity lately to avoid opioid adverse effects ranging from respiratory depression, postoperative ileus, sedation, nausea, vomiting and urinary retention.

Specific aims: The primary objective of this study is to compare blood pressure and heart rate between the fiberoptic and direct oral intubation using opioid free anesthesia induction. Secondary objectives include comparing the time needed for intubation and the incidence of postoperative sore throat, hoarseness, and upper airway trauma.

Methods: In this prospective randomized clinical trial, 90 (45 in each group) adults aging between 18 to 55 years, scheduled for elective surgery under general anesthesia, will be recruited over 1 year of work. Patients will be randomly allocated to 2 groups: The direct conventional laryngoscopy group performed with N3 (for females) or N4 (for males) Macintosh laryngoscope blade, and the fiberoptic guided intubation group.

Significance: Studies comparing hemodynamic stability using fiberoptic intubation versus direct oral intubation in opioid free anesthesia are limited. The present study will assess whether fiberoptic intubation causes less hemodynamic instability than direct oral intubation in opioid free anesthesia induction, which will benefit patients with normal airways.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status I and II
* Range age of 18-55 years' old
* Scheduled for elective surgery under general anesthesia.

Exclusion Criteria:

* History of cardiovascular diseases.
* History of lung disease.
* Hypertensive patient (BP> 140/90)
* Patient taking medications that affect blood pressure and heart rate
* Morbid obesity (BMI >30)
* Severe GERD
* Predicted difficult airway (Short TMD <6 cm, Upper li bite test grade III, Mallampati score

  >III)
* Neck instability
* Patient planned to receive rapid sequence intubation
* Patient refusal to participate
* History of difficult intubation/ ventilation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-09-11 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate | baseline and up to 5 mins upon intubation
  Heart rate (bpm)
Blood pressure | baseline and up to 5 mins upon intubation
  Blood pressure (mm Hg)

SECONDARY OUTCOMES:
time needed for intubation | between face mask removal and first ETCO2 reading in minutes
  time (between face mask removal and first ETCO2 reading in minutes)
incidence of postoperative sore throat | after 24 hrs
  Sore throat pain (0-10)
incidence of upper airway trauma | during intubation
  incidence of upper airway trauma (Yes or No)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Rouphael, MD, Principal Investigator — American University of Beirut Medical Center
Locations (1):
- Christian Rouphael, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No